CLINICAL TRIAL: NCT07073534
Title: Phase I/II Clinical Study on the Tolerability, Safety and Efficacy of SHR-1501 Combined With Adbelizumab in Patients With Malignant Tumors
Brief Title: Phase I/II Clinical Study of SHR-1501 Combined With Adbelizumab in Patients With Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1501-202
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: Patients With Advanced or Metastatic Malignant Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the combination of SHR-1501 and Adebrelimab (Experimental)
  Interventions: Drug: SHR-1501, Adebrelimab

INTERVENTIONS:
Drug: SHR-1501, Adebrelimab — the combination of SHR-1501 and Adebrelimab

SUMMARY:
This study is an open, multicenter phase I/II clinical study. The entire study is divided into three stages: dose escalation, dose expansion, and efficacy expansion. Objective: To evaluate the objective response rate (ORR), safety and tolerability of the combination of SHR-1501 and adibelizumab in the treatment of advanced malignant tumors, and to provide the recommended dose (RP2D) for subsequent clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical study, understand the research procedures and be able to sign the informed consent form in person.
2. Age: 18 to 75 years old (including both ends), gender not limited.
3. Subjects with locally advanced or metastatic solid tumors that have been histologically or cytologically confirmed to be inoperable for radical surgery or radical chemoradiotherapy, whose disease progresses after standard treatment, or who have no standard treatment plan, or are not suitable for standard treatment.
4. According to the efficacy evaluation criteria for Solid tumors (RECIST 1.1), there is at least one measurable lesion;
5. The ECOG physical condition score is 0 or 1.
6. The expected survival time is more than 3 months;

Exclusion Criteria:

1. Symptomatic or active central nervous system (CNS) tumor metastasis;
2. Other malignant tumors within five years before the first use of study drugs;
3. Uncontrolled tumor-related pain judged by the investigator;
4. Severe cardiovascular and cerebrovascular diseases;
5. Significant clinical bleeding symptoms within 3 months before the first study drug, and obvious fresh hemoptysis within 1 month before the first study drug;
6. Uncontrollable pleural effusion and/or ascites judged by the study or pleural effusion and/or ascites requiring intervention within 7 days before the first treatment
7. History of idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-related pneumonia requiring steroid therapy;,or active pneumonia at screening; or other moderate to severe pulmonary diseases that significantly affect pulmonary function;
8. Severe infection within 4 weeks before the start of study treatment
9. History of immunodeficiency
10. Used corticosteroids (>10 mg/day prednisone or equivalent) or other systemic immunosuppressants within 14 days before the first study drug.
11. Patients with active pulmonary tuberculosis infection within 1 year before enrollment as determined by medical history or imaging examination, or patients with a history of active pulmonary tuberculosis infection more than 1 year ago but without formal treatment
12. Patients whose adverse events caused by previous treatment have not recovered to ≤CTCAE grade 1
13. Patients whose previous treatment washout does not meet the following requirements: Patients who have received chemotherapy, biological therapy, targeted therapy, immunotherapy, or other unlisted clinical research drugs and other anti-tumor treatments within 4 weeks before the first use of the study drug
14. Patients who have experienced CTCAE grade 4 or grade 3 immune-related adverse events lasting for 4 weeks or longer after previous use of immune checkpoint inhibitors, or immune-related adverse events that led to treatment discontinuation, are not eligible for enrollment in this study.
15. Patients who have received >30 Gy chest radiotherapy within 24 weeks before the first use of the study drug, patients who have received >30 Gy non-chest radiotherapy within 4 weeks before the first use of the drug (subjects who have completed brain metastasis radiotherapy 14 days before the first use of the drug can be enrolled), and patients who have received ≤30 Gy within 14 days before the first use of the drug Gy of palliative radiation;
16. Subjects who have undergone surgery on important organs (excluding puncture biopsy) within 4 weeks before the first use of the study drug, have had significant trauma, or need to undergo elective surgery during the trial;
17. Active, known or suspected autoimmune diseases and history of autoimmune diseases.
18. Using attenuated live vaccines within 28 days before the first use of the study drug, or anticipating the need to use attenuated live vaccines during the study treatment;
19. Pregnant or lactating women or female subjects who plan to become pregnant during the study and within 6 months after the last use of the study drug;
20. Those who are known to be allergic to any component or excipient of the study drug; or have a history of severe allergic reactions to other monoclonal antibodies/fusion protein drugs;
21. The investigators judge that the subjects have other factors that may affect the study results or force the termination of this study, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment, serious abnormal laboratory test values, family or social factors, and other situations that may affect the safety of the subjects or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 21 Days or 28 days
  evaluate the safety in the doses escalation
Maximum tolerated dose or Maximum-administered dose | Approximately 1 years
  evaluate the safety in the doses escalation
Recommended Phase 2 dose (RP2D) | Approximately 2years.
  evaluate the safety and curative effect in the doses escalation
Objective response rate(ORR) | Approximately 2 years
  Preliminary evaluation of the effectiveness of the combination of SHR-1501 and Adebrelimab
The incidence and severity of adverse events (AE)/serious adverse events (SAE) (rated based on CTCAE v5.0) | 21 Days，Approximately 2 years
  Preliminary safety of the effectiveness of the combination of SHR-1501 and Adebrelimab

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of SHR-1501 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of the combination of SHR-1501 and Adebrelimab
Time to maximum concentration (Tmax) of SHR-1501 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of the combination of SHR-1501 and Adebrelimab
Areas under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of SHR-1501 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of the combination of SHR-1501 and Adebrelimab
Steady-state valley concentration (Cmin)of SHR-1501 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of Steady-state valley concentration
Accumulation ratio（Rac） of SHR-1501 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of the combination of SHR-1501 and Adebrelimab
Anti-drug antibody of SHR-1501 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of the combination of SHR-1501 and Adebrelimab
Duration of response(DoR) | Approximately 2 years
  Preliminary evaluation of the effectiveness of the combination of SHR-1501 and Adebrelimab
Disease control rate （DCR） | Approximately 2 years
  Preliminary evaluation of the effectiveness of the combination of SHR-1501 and Adebrelimab
Progression free survival （PFS ） | Approximately 2 years
  Preliminary evaluation of the combination of SHR-1501 and Adebrelimab
Overall survival（OS） | Approximately 2 years
  Preliminary evaluation of the effectiveness of the combination of SHR-1501 and Adebrelimab

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided